CLINICAL TRIAL: NCT04940741
Title: Proof of Efficacy, Maintenance of Efficacy, Long-term Safety and Investigation of the Potential for Dependence and Abuse and the Effect of Abrupt Drug Withdrawal of VER-01 in the Treatment of Patients With Chronic Non-specific Low Back Pain
Brief Title: Efficacy and Safety of VER-01 in the Treatment of Patients With Chronic Non-specific Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertanical GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VER-CLBP-001
Record Dates: First submitted 2021-06-07; First posted 2021-06-28 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Chronic Non-specific Low Back Pain

STUDY DESIGN:
Intervention Model Description: Phase A: randomised, double-blind, placebo-controlled (Efficacy and safety) Phase B: Open-label treatment (long-term safety) Phase C: Open-label treatment (long-term safety) Phase D: randomised, double-blind, placebo-controlled (maintenance of efficacy)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: different phases: open-label treatment and randomised, double-blind, placebo-controlled treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VER-01 (Experimental): VER-01 is administered orally (b.i.d.) using a dosing syringe. One unit corresponds to 2.5 mg THC. The optimal dose is titrated on a patient-by-patient basis. The maximum daily dose should not exceed 13 dose units (32.5 mg THC).
  Interventions: Drug: VER-01
- Placebo (Placebo Comparator): The Placebo is administered orally (b.i.d.) using a dosing syringe. The optimal dose is titrated on a patient-by-patient basis, analogous to VER-01.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VER-01 — standardised cannabis extract (containing 21 mg THC per gram drug product)
  Arms: VER-01
Other: Placebo — comparator without active ingredient
  Arms: Placebo

SUMMARY:
Analysis of the efficacy, maintenance of efficacy, long-term safety, and investigation of the potential for dependence and abuse and the effect of abrupt drug withdrawal of VER-01 in the treatment of patients with chronic non-specific low back pain when drug treatment is indicated and previous optimised treatments with non-opioid analgesics have not led to sufficient pain relief or were unsuitable due to contraindications or intolerance.

DETAILED DESCRIPTION:
The study is divided into four phases: Phase A, B, C and D. All patients who have completed Phase A and for whom the investigator considers further participation to be safe shall begin Phase B. Phases C and D run in parallel, so that patients who have completed Phase B and for whom the investigator considers further participation to be safe can be assigned to one of the two phases.

Phases A and D follow a double-blind, placebo-controlled design, while Phase B and C have an open-label design.

The main goal of Phase A is to demonstrate the efficacy of VER-01 compared to placebo. In Phase B and C the main goal is the investigation of long-term safety of VER-01. In Phase D the primary objective is to demonstrate the maintenance of efficacy of VER-01 on a placebo-controlled basis.

The potential for dependence and abuse will be analyzed in all Phases (A,B,C,D), while the effect of abrupt drug withdrawal of VER-01 will be analyzed in Phase C and D.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients (18 years and older)
2. Chronic (for at least three months) non-specific pain in the lower back (between the lower ribcage and the gluteal folds)
3. Pain intensity on average at least 4 points on an 11-point NRS (one month before the start of the study)
4. Patients with indicated drug treatment where previous optimised treatments with non-opioid analgesics have not led to sufficient pain relief or were unsuitable due to contraindications or intolerance.
5. Willingness of both men and women to use a reliable method of contraception during study participation and for three months after taking the last dose of the IMP
6. Signed patient information and informed consent form is available
7. Understanding of the German language, ability to give consent and compliance
8. The patient has understood the instructions to avoid changes in lifestyle and dietary habits
9. The patient has understood the principle of the patient diary and gives their consent to keep it as instructed

Additional for Phase A

a1. Pain intensity averaged at least 4 points on an 11-point NRS (there must be at least 5 pain intensity readings in the morning from the run-in phase)

a2. Willingness not to take any analgesic medication (non-opioid and opioid analgesics as well as adjuvant analgesics) during participation in study Phase A (except rescue medication)

a3. Willingness to continue a current non-drug therapy unchanged as planned during participation in Phase A

Additional for Phase B

b1. Previous and complete participation in Phase A until and including Visit A6

b2. Patient wishes to participate voluntarily in the long-term study

b3. From the investigator's point of view, further participation is considered medically safe

b4. Willingness not to take any additional analgesic medication (non-opioid and opioid analgesics as well as adjuvant analgesics) during the last three weeks of study Phase B (except rescue medication).

Additional for Phase C

c1. Previous and complete participation in Phase B until and including Visit B10

c2. Patient wishes to participate voluntarily in the long-term study

c3. From the investigator's point of view, further participation is considered medically safe

Additional for Phase D

d1. Previous and complete participation in Phase B until and including Visit B10 (patients received Ver-01 for 26 weeks)

d2. Patient has experienced a pain score improvement of at least 30% in treatment Phase B (mean value of the study week 43 compared to the mean value of the run-in phase, there must be at least four values from study week 43 and five values from the run-in phase)

d3. Patient wishes to participate voluntarily in the study

d4. From the investigator's point of view, further participation is considered medically safe

d5. Willingness not to take any analgesic medication (non-opioid and opioid analgesics as well as adjuvant analgesics) during participation in study Phase D (except rescue medication)

d6. Willingness to continue a current non-drug therapy unchanged as planned during study

Exclusion Criteria:

1. Professional groups for which the ability to operate machinery and drive vehicles is the primary activity (including truck, bus and forklift drivers, pilots)
2. Alcohol/drug/medication abuse and previous or current intake of methadone in the patient's medical history or suspected by the investigator
3. Intake of analgesic medication (non-opioid and opioid analgesics as well as adjuvant analgesics) within seven days prior to the start of the study
4. Taking cannabis-based products within 30 days prior to the start of the study
5. HIV, dementia (which impairs the assessment of symptoms)
6. Severe forms of the following diseases: Anaemia,hematological/autoimmune/endocrinal/ renal/hepatic/respiratory/cardiovascular or gastrointestinal diseases, symptomatic peripheral vascular diseases
7. Cardiovascular event in the past three months, poorly managed high blood pressure, untreated hypothyroidism, patients with Crigler-Najjar syndrome or Rotor syndrome, surgery within the past two months
8. Severe mental illnesses (e.g. psychosis, schizophrenia, bipolar disorder), severe depression that is not due to the chronic non-specific low back pain, or individuals at risk of suicide (examined using the MINI questionnaire)
9. Severe mental illness (psychosis, schizophrenia, bipolar disorder, severe depression, anxiety disorder) in a first-degree relative (parents and children); suicide in a first-degree relative (parents and children)
10. Patients with an active cancer or tumor-related pain or severe pain due to physical injury
11. Other painful comorbidities, excluding low back pain, that could interfere with the patient's evaluation during the study or the assessment of pain
12. Well-known strong adverse events in connection with cannabis consumption before the start of the study
13. Known allergy to cannabis and/or sesame seeds and products derived from them
14. Known hypersensitivity to the ingredients of the rescue medication
15. Planned blood donation, planned sperm or egg donation, planned freezing of eggs or sperm
16. Pregnancy, breastfeeding, desire to have children (within the next 20 months)
17. Participation in another clinical trial within the past 30 days before the start of the study
18. Inability to give consent, care dependency, patient has a legal guardian/caregiver, or is immobile
19. The patient is in need of special protection (e.g., incarcerated; institutionalized by a court or judicial authority; in a dependent or employment relationship with the sponsor, an external service provider of the sponsor (who is involved in the study conduct), the investigator, or the study site).

Additional for Phase A:

a1. In the case of a current non-drug therapy (e.g. physical or behavioural therapy, acupuncture,massage, thermotherapy), which significantly modulates the perception of pain, it was not maintained unchanged for at least eight weeks prior to study participation in Phase A.

Additional for Phase D

d1. Intake of additional analgesic medication (non-opioid and opioid analgesics as well as adjuvant analgesics) within 21 days prior to the start of study Phase D (except rescue medication).

d2. In the case of a current non-drug therapy (e.g. physical or behavioural therapy, acupuncture,massage, thermotherapy) that significantly modulates the perception of pain, it was not maintained unchanged for at least nine weeks prior to the start of study Phase D.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Phase A: Efficacy based on pain reduction | Baseline up to 15 weeks
  Change in average pain intensity compared to baseline on an 11-point Numerical Rating Scale (NRS, where 0=no pain to 10=worst pain imaginable) (mean value of study week 15 compared to the mean value of the seven-day run-in phase with daily documentation of pain intensity in the morning).
Phase B: Safety based on occurrence of treatment-related AEs/SAEs | Up to 29 weeks
  Safety and adverse reactions based on occurrence of treatment-related AEs/SAEs
Phase C: Safety based on occurrence of treatment-related AEs/SAEs | Up to 28 weeks
  Safety and adverse reactions based on occurrence of treatment-related AEs/SAEs
Phase D: Maintenance of efficacy | Up to 4 weeks (from date of randomization R2 until the first day of treatment failure)
  Time until treatment failure defined as the time in days from randomization to phase D (R2) until the first day of treatment failure. Treatment failure is assessed by the daily calculated seven-day mean value of the pain score (11 point Numerical Rating Scale, NRS, where 0=no pain to 10=worst pain imaginable) in the morning during the treatment period, which must have deteriorated by at least 20% and at least one point compared to baseline (mean value of study week 43). The first day of treatment failure is then the earliest day within this seven-day time window to which this criterion applies as a single day. Furthermore, treatment failure is defined as a premature discontinuation of treatment for selected reasons.

SECONDARY OUTCOMES:
Phase A, B, C, D: Mean change in neuropathic pain | Day 1, day 106, day 309, day 351, day 505
  Absolute change compared to baseline (day1) Neuropathic Pain Symptom Inventory (NPSI) total score at the end of each treatment phase in patients with neuropathic pain
Phase A, B, C, D: Change in pain intensity in the morning, as well as in the morning and evening | Baseline up to 72 weeks
  Absolute changes from baseline in mean pain intensity at the end of each treatment phase measured in the morning (primary endpoint of Phase A) or morning and evening on an 11-point Numerical Rating Scale (NRS, where 0=no pain to 10=worst pain imaginable)
Phases A, B, C and D: Pain responders (30 percent and 50 percent) in the morning, as well as in the morning and evening | Baseline up to 72 weeks
  The number and proportion of 30 percent and 50 percent pain responders in the morning, and morning and evening at the end of each treatment phase.
Phases A, B, C and D: Sleep quality (NRS) | Baseline up to 72 weeks
  The absolute change from baseline in mean sleep quality at the end of each treatment phase measured on an 11-point Numerical Rating Scale (NRS, where 0=not impacted to 10=completely impacted)
Phase A: Sleep quality (MOS-SS) | Day 1, Day 22, Day 50, Day 78, Day 106
  Absolute changes from baseline of sleep quality measured by Medical Outcomes Study Sleep Scale (MOS-SS) per survey point
Phase A: Intake of rescue and concomitant medication | Up to 16 weeks
  Cumulative dose of rescue medication taken in Phase A
Phase D: Intake of rescue and concomitant medication | Up to 6 weeks
  Cumulative dose of rescue medication taken in Phase D
Phases A, B, C and D: Depression Anxiety Stress Scales (DASS) | Baseline up to 72 weeks
  Scores and absolute changes from baseline of depression, anxiety and stress levels measured by the DASS (where 0=did not apply to me at all to 3=affected me very greatly or most of the time) per time point of assessment
Phases A, B, C and D: Global assessment of symptoms (patient global impression of change, PGIC) | Day 106, day 309, day 491, day 337
  Percentage of patients by category of the global assessment of symptoms (PGIC, 7-point Likert scale where 0=very much better to 6=very much worse) by the patient per survey point
Phases A, B, C and D: Satisfaction with the treatment result - patient | Day 106, day 309, day 491, day 337
  Percentage of patients by category of the satisfaction with the treatment outcome (5-point Likert scale, where 0=very satisfied to 4=very unsatisfied) by the patient per survey point
Phases A, B, C and D: Satisfaction with the treatment result - investigator | Day 106, day 309, day 491, day 337
  Percentage of patients by category of satisfaction with the treatment outcome (5-point Likert scale, where 0=very satisfied to 4=very unsatisfied) by the investigator per survey point.
Phases A, B, C and D: Satisfaction with tolerability - patient | Day 106, day 309, day 491, day 337
  Percentage of patients by category of satisfaction with the tolerability (5-point Likert scale, where 0=very satisfied to 4=very unsatisfied) by the patient per survey point
Phase A: Safety and adverse reactions | Up to 16 weeks
  Safety and adverse reactions based on occurrence of treatment-related AEs/SAEs
Phase D: Safety and adverse reactions | Up to 6 weeks
  Safety and adverse reactions based on occurrence of treatment-related AEs/SAEs
Phases A, B, C and D: Quality of life scores (Short Form 36, SF-36) | Day 1, day 22, day 50, day 78, day 106, day 309, day 491, day 337
  Scores in quality of life measured per survey point
Phases A, B, C and D: Quality of life absolute changes (Short Form 36, SF-36) | Day 1, day 22, day 50, day 78, day 106, day 309, day 491, day 337
  Absolute changes in quality of life from baseline (day 1) measured per survey point
Phase A: Scores in bodily function and impairment due to low back pain (Roland Morris Disability Questionnaire, RMD) | Day 1, day 22, day 106
  Scores in bodily function and impairment due to low back pain assessed by the RMD per survey point
Phase A: Absolute changes in bodily function and impairment due to low back pain(Roland Morris Disability Questionnaire, RMD) | Day 1, day 22, day 106
  Absolute changes in bodily function and impairment due to low back pain assessed by the RMD per survey point
Phases A, B, C and D: Addiction (Addiction Behaviors Checklist ,ABC) | Day 22, day 50, day 78, day 106, day 127, day 183, day 239, day 309, day 365, day 421, day 491, day 337
  The absolute number of positive answers of the ABC
Phase C: Diagnosis of substance dependence ICD-10 (International Statistical Classification of Diseases and Related Health Problems) | Day 491
  The absolute number of positive answers according to the German Bundesärztekammer (2007) is summarized descriptively according to the standard for continuous parameters.
Phase A, B, C and D: Adverse events (AEs) | Through study completion, up to 72 weeks
  Occurrence of AEs/SAEs
Phase C: Withdrawal symptoms (Cannabis Withdrawal Scale, CWS) | Up to 2 weeks
  Sum scores for intensity and functional impairment are descriptively analysed according to Allsop et al.
Phase D: Withdrawal symptoms (Cannabis Withdrawal Scale, CWS) | Up to 4 weeks
  Sum scores for intensity and functional impairment are descriptively analysed according to Allsop et al.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Nadstawek, Prof., Principal Investigator — Schmerzzentrum Bonn
Locations (1):
- Emovis GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karst M, Meissner W, Sator S, Kessler J, Schoder V, Hauser W. Full-spectrum extract from Cannabis sativa DKJ127 for chronic low back pain: a phase 3 randomized placebo-controlled trial. Nat Med. 2025 Dec;31(12):4189-4196. doi: 10.1038/s41591-025-03977-0. Epub 2025 Sep 29. PMID 41023483